CLINICAL TRIAL: NCT04828018
Title: Care of the Ageing Veteran Population: Developing an Evidence Base for the Royal Hospital Chelsea Model of Care
Status: Completed | Type: Observational
Sponsor: Northumbria University (Other)
Collaborators: Royal Hospital Chelsea (Unknown)
Responsible Party: Sponsor
Other Study IDs: 119967
Record Dates: First submitted 2021-03-02; First posted 2021-04-01 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Quality of Life; Aging Well

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Key Staff: Key Staff will take part in one interview lasting up to 60 minutes
  Interventions: Other: Coffee Morning; Other: Recruitment Leaflets; Other: Consent Form completion; Other: Participant Information Sheet; Other: Key Staff Interviews
- In-Pensioners: Royal Hospital Chelsea In-Pensioners will take part in one interview lasting up to 90 minutes and complete n=2 Quality of Life Questionnaires (ICECAP-A and WHOQOL-BREF) at the start of their qualitative interview.
  Interventions: Other: Coffee Morning; Other: Recruitment Leaflets; Other: Consent Form completion; Other: Participant Information Sheet; Other: In-Pensioner Resident Interviews; Other: ICECAP-A Quality of Life Questionnaire; Other: WHOQOL-BREF Quality of Life Questionnaire
- New In-Pensioner: New In-Pensioners wil be asked to complete a total of n=4 Quality of Life Questionnaires (ICECAP-A and WHOQOL-BREF), n=2 on admission to Royal Hospital Chelsea and n=2 six months after admission.
  Interventions: Other: New In-Pensioner Resident Information Pack; Other: ICECAP-A Quality of Life Questionnaire; Other: WHOQOL-BREF Quality of Life Questionnaire

INTERVENTIONS:
Other: Coffee Morning — Coffee mornings (a maximum of n=2) will be held to raise awareness of the project and to promote participant recruitment. These will be held remotely via video conference if Covid-19 restrictions prevent in-person attendance by the researcher.
  Groups: In-Pensioners; Key Staff
Other: Recruitment Leaflets — Recruitment leaflets will be hand-delivered to all In-Pensioner residents at Royal Hospital Chelsea. Leaflets will be delivered internally by Royal Hospital Chelsea internal mail-room
  Groups: In-Pensioners; Key Staff
Other: Consent Form completion — All participants will be asked to complete Consent Forms before engaging in the study. The researcher will be available to answer any questions via phone calls if required.
  Groups: In-Pensioners; Key Staff
Other: Participant Information Sheet — All participants will receive Information Sheets which they will read in their own rooms (or elsewhere for Key Staff). The researcher will be available to answer any questions via phone calls if required.
  Groups: In-Pensioners; Key Staff
Other: New In-Pensioner Resident Information Pack — New In-Pensioner resident information packs will be distributed by a member of RHC staff as part of their 'arrivals' process and six months after residency at RHC. The researcher will be available to answer any questions via phone calls if required.
  Groups: New In-Pensioner
Other: Key Staff Interviews — Key Staff interviews will take place with the Researcher in a private space at Royal Hospital Chelsea. If Covid-19 restrictions are in place, 'online' interviews will take place using a digital platform such as 'Skype', 'Teams' or 'Zoom'.
  Groups: Key Staff
Other: In-Pensioner Resident Interviews — In-Pensioner resident interviews will take place with the Researcher in a private space at Royal Hospital Chelsea. If Covid-19 restrictions are in place, 'online' interviews will take place using a digital platform such as 'Skype', 'Teams' or 'Zoom'.
  Groups: In-Pensioners
Other: ICECAP-A Quality of Life Questionnaire — New In-Pensioner residents and In-Pensioner residents taking part in the Qualitative Interviews will be asked to complete n=2 QoL questionnaires. New In-Pensioners will be asked to complete their QoL measures when the individual takes up residence at Royal Hospital Chelsea, the second six months later. In-Pensioner residents taking part in the interviews will be asked to complete the questionnaire at the start of the interview.
  Groups: In-Pensioners; New In-Pensioner
Other: WHOQOL-BREF Quality of Life Questionnaire — New In-Pensioner residents and In-Pensioner residents taking part in the Qualitative Interviews will be asked to complete n=2 QoL questionnaires. New In-Pensioners will be asked to complete their QoL measures when the individual takes up residence at Royal Hospital Chelsea, the second six months later. In-Pensioner residents taking part in the interviews will be asked to complete the questionnaire at the start of the interview.
  Groups: In-Pensioners; New In-Pensioner

SUMMARY:
Royal Hospital Chelsea (RHC) has provided a sheltered housing environment alongside integrated health and social care and comradeship for British Army veterans since 1692, following a decree by King Charles II to aid the "relief of veterans broken by age and war" (RHC, 2018). Today approximately 300 In-Pensioners, known globally as 'Chelsea Pensioners' live at RHC. They also have access to an on-site infirmary providing nursing or personal care for up to 68 people (CQC, 2019).

RHC is in central London (UK) and comprises of several historical buildings, protected by the organisations Mission Statement to "…safeguard their historic home for the veterans of tomorrow". In-Pensioner's must have served in the British Army as a non-commissioned officer (or have served at least 12 years 'in the ranks' prior to becoming a commissioned officer), be aged 65 or over, be free of any financial obligations to dependents, and at the time of admission be able to live independently. Traditionally a male-only residence, RHC welcomed its first female Army veteran in 2009.

There is an absence of evidence to support the impact of care delivery and the Chelsea Pensioner experience, with the only evidence being RHC Annual and Care Quality Commission (CQC) reports which focus on strategic and operational matters rather than the impact of the wider social care or environment.

This lack of evidence presents a unique opportunity to evaluate RHC's current service provision, inform future direction and address the hiatus in evidence-based research to quantify the impact of its model of care.

DETAILED DESCRIPTION:
The research will seek to address two main aims:

1. To gain an understanding of the current Royal Hospital Chelsea (RHC) model of care by:

   1. Evidencing the influence the model of care has on In-Pensioner health outcomes
   2. Understanding the influence the model of care has on wider social care provision
   3. Reflecting on the contribution the environment has on the In-Pensioner experience, their health outcomes, and quality of life
2. To inform future RHC care provision by:

   1. Mapping current services, future need and sustainability of the model
   2. Projecting findings to inform the growth of existing services for future generations of ageing veterans

The findings will inform RHC strategic direction as it continues to deliver care provision to current and future generations of veteran, identify the value of RHC interventions, and explore any development of service provision in the form of potential outreach care. Further, the findings will look to inform wider social care provision which may contribute to national health and social care policy.

The findings of the study may be applicable to the wider care provision within similar residential care establishments as they will seek to present service delivery findings from both a staff (care provider) and resident (care recipient) perspective and evidence best practice.

The findings may contribute to national health and social care policy (UK).

Key staff and Royal Hospital Chelsea 'In-Pensioner' residents will be interviewed for this study. New In-Pensioner residents will be invited to complete two Quality of Life Questionnaires (one on arrival and one six months later).

ELIGIBILITY:
Inclusion Criteria:

• Participants identified as Key Staff, In-Pensioner residents and new In-Pensioners at Royal Hospital Chelsea will be eligible to be included in the study.

Exclusion Criteria:

* Anyone who is not employed by Royal Hospital Chelsea and identified as a Key Member of staff, or is not an In-Pensioner resident at Royal Hospital Chelsea will be excluded from the study.
* Any potential participant who does not complete a consent form will be excluded from the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population comprises key staff employees of Royal Hospital Chelsea (n=19), residents of Royal Hospital Chelsea (known as In-Pensioners) (n=25) and new In-Pensioners (n=40)who are admitted to the institution over a 12 month period (to complete n=2 Quality of Life Questionnaires only)
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2024-01-24 (Actual)

PRIMARY OUTCOMES:
Key Staff Interviews | Interviews, lasting 60 minutes per interview, will take place over a 3-month period. Data analysis will take place over a 10-month period during years two and three of the study.
  Semi-structured 'in-person' interviews will take place with n=25 key staff at Royal Hospital Chelsea. Analysis of this data will be assessed using NVIVO software.
In-Pensioner Interviews | Interviews, lasting up to 90 minutes per interview, will take place over an 8-month period. Data analysis will take place over a 10-month period during years two and three of the study.
  Semi-structured 'in-person' interviews will take place with n=25 Royal Hospital Chelsea In-Pensioner residents. Analysis of this data will be assessed using NVIVO software.
Royal Hospital Chelsea Documentation Review | Documentation review and data analysis will take place ahead of the writing-up phase of the study, approximately 15 months.
  Royal Hospital Chelsea documents including organisational policies, annual reports, healthcare governance reports and data from the Margaret Thatcher Infirmary will be reviewed. Data collected will be analysed using SPSS software.
ICECAP-A Quality of Life Questionnaire | Questionnaires will be completed over a 12-month period during years two and three of the study. Data analysis will take place over a 10-month period during years two and three of the study.
  The ICECAP-A Quality of Life questionnaire will be completed by new In-Pensioner residents, and In-Pensioners selected for Qualitative Interview at Royal Hospital Chelsea. Data analysis will take place using SPSS software.
  ICECAP-A is the ICEpop CAPability measure for Adults Quality of Life measure and is scored using the Likert Scale framework. The questionnaire has a minimum value of 1 and a maximum value of 4, with the maximum value indicating a better outcome.
WHOQOL-BREF Quality of Life Questionnaire | Questionnaires will be completed over a 12-month period during years two and three of the study. Data analysis will take place over a 10-month period during years two and three of the study.
  The WHOQOL-BREF Quality of Life questionnaire will be completed by new In-Pensioner residents, and In-Pensioners selected for Qualitative Interview at Royal Hospital Chelsea. Data analysis will take place using SPSS software.
  The WHOQOL-BREF is the World Health Organisation Quality of Life - Brief questionnaire which is a short-form version of the WHOQOL-100 Quality of Life measure and is scored using the Likert Scale framework. The questionnaire has a minimum value of 1 and a maximum value of 5, with the maximum value indicating a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Gemma Wilson-Menzfeld, PhD, Principal Investigator — Northumbria University
Locations (1):
- Royal Hospital Chelsea, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Currently in discussion